CLINICAL TRIAL: NCT06252259
Title: Choose to Move (CTM): Implementation and Impact Evaluation of an Adapted Health-Promoting Program for Equity-Deserving Older Adults
Brief Title: Evaluating Implementation and Impact of the Adapted Choose to Move (CTM) Program
Acronym: CTM
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Active Aging Society (Other)
Responsible Party: Principal Investigator, Heather McKay, Professor, University of British Columbia
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H22-03385; HG2-185013 (Other Grant/Funding Number: Canadian Institutes of Health Research)
Record Dates: First submitted 2024-02-01; First posted 2024-02-09 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Aging; Mobility Limitation; Physical Inactivity; Sedentary Behavior; Loneliness; Social Isolation
Keywords: Older adults; Physical activity; Mobility; Social isolation; Loneliness; Social connectedness; Behavior change; Implementation; Implementation strategy; Health equity; Adaptation; Readiness; Feasibility; Acceptability; Dose; Fidelity; Effectiveness
MeSH Terms: conditions — Mobility Limitation; Sedentary Behavior; Social Isolation; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Ethnicity and Culture in Focus (Experimental): CTM (Phase 5) is a 3-month, flexible, choice-based health-promoting program for low active older adults that can be delivered in-person or online. The program includes:
  * 1-on-1 Consultation: Participants meet 1-on-1 with their activity coach at the start of the program to set goals and develop a physical activity action plan tailored to their abilities, interests and resources. Older adults can choose to participate in individual or group-based activities.
  * Group Meetings: Participants will attend eight, 1-hour group-based meetings (max of 15 participants) led by their activity coach. Meetings cover a health-related discussion topic and provide time and space for social connection among participants. Meetings can be held online or in-person.
  The CTM program will be adapted for South Asian older adults, and may include additional intervention components customized for this population.
  Interventions: Behavioral: Choose to Move
- Men on the Move (Experimental): CTM (Phase 5) is a 3-month, flexible, choice-based health-promoting program for low active older adults that can be delivered in-person or online. The program includes:
  * 1-on-1 Consultation: Participants meet 1-on-1 with their activity coach at the start of the program to set goals and develop a physical activity action plan tailored to their abilities, interests and resources. Older adults can choose to participate in individual or group-based activities.
  * Group Meetings: Participants will attend eight, 1-hour group-based meetings (max of 15 participants) led by their activity coach. Meetings cover a health-related discussion topic and provide time and space for social connection among participants. Meetings can be held online or in-person.
  The CTM program will be adapted for older men, and may include additional intervention components customized for this population.
  Interventions: Behavioral: Choose to Move
- The Forgotten North (Experimental): CTM (Phase 5) is a 3-month, flexible, choice-based health-promoting program for low active older adults that can be delivered in-person or online. The program includes:
  * 1-on-1 Consultation: Participants meet 1-on-1 with their activity coach at the start of the program to set goals and develop a physical activity action plan tailored to their abilities, interests and resources. Older adults can choose to participate in individual or group-based activities.
  * Group Meetings: Participants will attend eight, 1-hour group-based meetings (max of 15 participants) led by their activity coach. Meetings cover a health-related discussion topic and provide time and space for social connection among participants. Meetings can be held online or in-person.
  The CTM program will be adapted for older adults living in Northern BC, and may include additional intervention components customized for this population.
  Interventions: Behavioral: Choose to Move

INTERVENTIONS:
Behavioral: Choose to Move — As described under study arm description

SUMMARY:
Choose to Move (CTM) is a 3-month, choice-based health-promoting program for low active older adults being scaled-up across British Columbia (BC), Canada. In Phase 5, the goal of CTM is to enhance physical activity, mobility and social connectedness in three target populations: South Asian older adults, older men, and older adults living in Northern BC. To do so, the investigators will support community-based seniors' services (CBSS) organizations through a readiness-building process so they can adapt CTM and deliver the program to these populations.

This study has two main research questions:

1. How are adapted CTM programs delivered ('implementation outcomes') and what factors influence delivery ('implementation determinants')?
2. What is the impact of the adapted CTM programs on health outcomes of older adults?

DETAILED DESCRIPTION:
Choose to Move (CTM) a 3-month, choice-based health-promoting program for low active older adults being scaled-up in phases across British Columbia (BC), Canada. To date (Phases 1-4), CTM participants have included mostly white older women living in large urban centres. In Phase 5, the investigators aim to expand the reach of CTM to three target populations: South Asian older adults, older men, and older adults living in Northern BC.

Within CTM (Phase 5), trained activity coaches support older adults in two ways. First, in a one-on-one consultation, activity coaches help participants to set goals and create action plans for physical activity tailored to each person's interests and abilities. Older adults can choose to participate in individual or group-based activities. Second, activity coaches facilitate 8 group meetings with small groups of participants.

In this study, the central support unit (CSU) will work with community-based seniors' services (CBSS) organizations to adapt CTM to 'best fit' these target populations of older adults, and build capacity in these organizations to deliver CTM. The investigators will then evaluate the implementation of the adapted programs, and the impact of the adapted programs on older adults' physical and social health.

Objectives:

1. To assess whether CTM (Phase 5) was implemented as planned (fidelity) and investigate factors that support or inhibit its implementation at scale (Part I - Implementation Evaluation).
2. To assess the impact (effectiveness) of CTM (Phase 5) on the physical activity, mobility, and social connectedness of older adult participants (Part II - Impact Evaluation).
3. To assess whether participant-level benefits of CTM (Phase 5) are maintained 12 months after participants complete the CTM program.

Study Design:

The investigators use a hybrid type 2 effectiveness-implementation (Curran et al. 2012) pre-post study design to evaluate CTM Phase 5. The investigators use mixed methods (quantitative and qualitative) and collect data at 0 (baseline), 3 (post-intervention) and 15 (12-months post intervention) months to assess implementation and impact of CTM.

ELIGIBILITY:
Inclusion criteria:

* Central support unit staff member;
* Delivery partner organization staff member;
* Activity coach hired by delivery partner organization (activity coaches must speak English to participate in the evaluation);
* English-speaking older adults (aged >=50 years) who participate in CTM (recruited by delivery partner organizations) will be invited to participate in the evaluation;
* Punjabi-speaking older adults will also be invited to participate in the evaluation if they can read English or Punjabi and/or if the activity coach or a member of the research team has the necessary language skills to ensure effective communication of the Punjabi language translated consent form and surveys.

Exclusion criteria:

* non-English speaking delivery partner staff member
* non-English speaking activity coach

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 336 (Estimated)
Dates: Start 2024-08-06 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Change in physical activity | 0, 3, 15 months
  The single item physical activity questionnaire will be used to measure physical activity. Output variable is self-reported number of days/week ≥30 min physical activity in the past week (range 0-7).

SECONDARY OUTCOMES:
Change in capacity for mobility | 0, 3, 15 months
  Two items will assess participants' ability to walk a quarter of a mile and up 10 steps. The output variable is self- reported presence of mobility-disability (no/any difficulty walking 400m or climbing one flight of stairs).
Change in physical functioning | 0, 3, 15 months
  The Physical Functioning Subscale of the SF-36 will be used to assess the physical function aspect of mobility. The measure asks participants to rate if their health limits them in performing 10 different activities. The output variable is an average score (range 0-100) of physical functioning, where a higher score indicates a more favourable health state.
Change in loneliness | 0, 3, 15 months
  The three-item loneliness scale will be used to assess loneliness. Participants rate three aspects of loneliness. The output variable is loneliness score (range 3-9); lower scores indicate lower levels of loneliness.
Change in social isolation | 0, 3, 15 months
  A four-item questionnaire adapted from two questions on social contact frequency will be used to assess social isolation. The output variable is social isolation score (range 0-20); higher scores indicate lower levels of social isolation.
Change in social network | 0, 3, 15 months
  A six-item questionnaire will be used to assess social network. The output variable is an equally weighted sum (range 0-30) where higher scores indicate more social engagement.
Change in social connectedness | 0, 3, 15 months
  A single item will be used to assess sense of belonging as an indicator of social connectedness. The output variable is sense of belonging score (range 1-4) where lower scores indicate a stronger sense of belonging.
Change in health-related quality of life (EQ-5D-5L Profile) | 0, 3, 15 months
  The EQ-5D-5L consists of five dimensions (mobility, self-care, usual activities, pain/discomfort and anxiety/depression). Participants are asked to indicate their level of functioning (from 1 "no problems" to 5 "extreme problems") on each of the five dimensions of the EQ-5D-5L. The EQ-5D-5 L describes 3125 distinct health states, with 11111 representing the best and 55555 the worst possible health states. The investigators apply the Canadian EQ-5D-5 L scoring algorithm to generate index scores, which ranged from - 0.148 for the worst (55555) to 0.949 for the best (11111) health states.
Change in health-related quality of life (EQ-5D-5L Visual Analogue Scale) | 0, 3, 15 months
  Health status will be assessed with the EQ-5D-5L visual analogue scale. Participants report on their health on a visual analogue scale from 0 (worst health) to 100 (best health).
Change in physical activity (objective) | 0, 3, 15 months
  Physical activity will be assessed by accelerometers (worn for 7 days) in a subset of participants in the Men on the Move study arm. The output variables are minutes per day of light, moderate and vigorous physical activity.

OTHER OUTCOMES:
Reach-individual | 3 months
  Number of organizations and older adults participating in adapted CTM programs will be obtained from program records.
Reach-regional | 0 months
  The neighbourhood characteristics of the regions where CTM programs were delivered will be determined using the Canadian Social Environment Topology (CanSET) tool.
Context - CTM program (interview) | 3 months
  Aspects of the larger social, political and economic environment that may influence delivery of the adapted CTM program will be assessed by interview.
Acceptability - CTM program (survey) | 3 months
  DPOs perception that the adapted CTM program is agreeable or satisfactory will be assessed by survey (4 items each on a 1-5 Likert scale with 1 being completely disagree and 5 being completely agree; developed in house).
Adaptability - CTM program (survey) | 3 months
  Extent to which the adapted CTM program can be adapted, tailored, refined, or reinvented to meet local needs will be assessed by survey (4 items each on a 1-5 Likert scale with 1 being completely disagree and 5 being completely agree; developed in house).
Feasibility - CTM program (survey) | 3 months
  DPOs perception that the adapted CTM program can be successfully used within the organization will be assessed by survey (4 items each on a 1-5 Likert scale with 1 being completely disagree and 5 being completely agree; developed in house).
Appropriateness - CTM program (survey) | 3 months
  Extent to which the adapted CTM program fits with the mission, priorities, and values of organizations or setting will be assessed by survey (4 items each on a 1-5 Likert scale with 1 being completely disagree and 5 being completely agree; developed in house).
Cost - CTM program | 3 months
  Program delivery costs will be recorded using a cost capture template developed in house.
Culture - CTM program (interview) | 3 months
  DPOs' norms, values, and basic assumptions around selected health outcomes (physical activity, mobility, social health) will be assessed by interview with DPO staff.
Complexity- CTM program (interview) | 3 months
  Perceptions among the DPOs that the adapted CTM program is relatively difficult to understand and use; number of different intervention components will be assessed by interview with DPO staff.
Self-efficacy - CTM program (interview) | 3 months
  DPOs belief in their own capability to execute courses of action to achieve implementation goal will be assessed by interview with DPO staff.
Readiness (survey) | 0 months
  The extent to which an organization is both willing and able to implement a particular innovation will be assessed using a modified version of the Readiness Diagnostic Scale. This scale evaluates three components of readiness: motivation (14 items), general capacity (24 items), and innovation capacity (12 items). Each item is scored on a 1-7 Likert scale with 1 being Strongly Disagree and 7 being Strongly Agree.
Adoption - CTM program | 3 months
  Number of activity coaches trained to deliver the CTM program will be obtained from program records.
Dose delivered - CTM program (survey) | 3 months
  Number of group meetings (0-8) delivered by activity coaches will be assessed by survey (developed in house).
Fidelity - CTM program (survey) | 3 months
  Fidelity to planned delivery will be assessed via survey (designed in house) for activity coaches and older adult participants. Higher scores (1-5 Likert scale) indicate better adherence to planned delivery.
Fidelity - CTM program (interview) | 3 months
  Fidelity to planned delivery will be assessed via interview with activity coaches and older adult participants.
Participant Responsiveness - CTM program (survey) | 3 months
  Program satisfaction will be assessed via participant (older adults) survey (designed in house). Higher scores (1-5 Likert scale) indicate higher participant satisfaction with the intervention.
Participant Responsiveness - CTM program (interview) | 3 months
  Program satisfaction will be assessed via interview with older adult CTM participants.
Adaptation - CTM program (survey) | 3 months
  Planned or purposeful changes to the delivery of the adapted CTM program by activity coaches will be assessed by survey (short answer responses; developed in house). Coaches will indicate if they made any adaptations to the program (yes/no) and to provide details of any adaptations such as why it needed to occur.
Adaptation - CTM program (interview) | 3 months
  Planned or purposeful changes to the delivery of the adapted CTM program by activity coaches will be assessed by interview.

CONTACTS AND LOCATIONS:
Overall Officials: Heather A McKay, PhD, Principal Investigator — University of British Columbia; Joanie Sims Gould, PhD, Principal Investigator — University of British Columbia; Dawn Mackey, PhD, Principal Investigator — Simon Fraser University; Farinaz Havaei, RN, PhD, Principal Investigator — University of British Columbia
Locations (1):
- Active Aging Research Team, Robert H. N. Ho Research Centre, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Curran GM, Bauer M, Mittman B, Pyne JM, Stetler C. Effectiveness-implementation hybrid designs: combining elements of clinical effectiveness and implementation research to enhance public health impact. Med Care. 2012 Mar;50(3):217-26. doi: 10.1097/MLR.0b013e3182408812. PMID 22310560
- [Background] Milton K, Bull FC, Bauman A. Reliability and validity testing of a single-item physical activity measure. Br J Sports Med. 2011 Mar;45(3):203-8. doi: 10.1136/bjsm.2009.068395. Epub 2010 May 19. PMID 20484314
- [Background] Hughes ME, Waite LJ, Hawkley LC, Cacioppo JT. A Short Scale for Measuring Loneliness in Large Surveys: Results From Two Population-Based Studies. Res Aging. 2004;26(6):655-672. doi: 10.1177/0164027504268574. PMID 18504506
- [Background] Macdonald HM, Nettlefold L, Bauman A, Sims-Gould J, McKay HA. Pragmatic Evaluation of Older Adults' Physical Activity in Scale-Up Studies: Is the Single-Item Measure a Reasonable Option? J Aging Phys Act. 2022 Feb 1;30(1):25-32. doi: 10.1123/japa.2020-0412. Epub 2021 Aug 4. PMID 34348228
- [Background] Simonsick EM, Newman AB, Visser M, Goodpaster B, Kritchevsky SB, Rubin S, Nevitt MC, Harris TB; Health, Aging and Body Composition Study. Mobility limitation in self-described well-functioning older adults: importance of endurance walk testing. J Gerontol A Biol Sci Med Sci. 2008 Aug;63(8):841-7. doi: 10.1093/gerona/63.8.841. PMID 18772472
- [Background] Veroff JB. The dynamics of help-seeking in men and women: a national survey study. Psychiatry. 1981 Aug;44(3):189-200. PMID 7267859
- [Background] Bauer GR, Braimoh J, Scheim AI, Dharma C. Transgender-inclusive measures of sex/gender for population surveys: Mixed-methods evaluation and recommendations. PLoS One. 2017 May 25;12(5):e0178043. doi: 10.1371/journal.pone.0178043. eCollection 2017. PMID 28542498
- [Background] Ware JE Jr, Sherbourne CD. The MOS 36-item short-form health survey (SF-36). I. Conceptual framework and item selection. Med Care. 1992 Jun;30(6):473-83. PMID 1593914
- [Background] Proctor E, Silmere H, Raghavan R, Hovmand P, Aarons G, Bunger A, Griffey R, Hensley M. Outcomes for implementation research: conceptual distinctions, measurement challenges, and research agenda. Adm Policy Ment Health. 2011 Mar;38(2):65-76. doi: 10.1007/s10488-010-0319-7. PMID 20957426
- [Background] McKay H, Naylor PJ, Lau E, Gray SM, Wolfenden L, Milat A, Bauman A, Race D, Nettlefold L, Sims-Gould J. Implementation and scale-up of physical activity and behavioural nutrition interventions: an evaluation roadmap. Int J Behav Nutr Phys Act. 2019 Nov 7;16(1):102. doi: 10.1186/s12966-019-0868-4. PMID 31699095
- [Background] Durlak JA, DuPre EP. Implementation matters: a review of research on the influence of implementation on program outcomes and the factors affecting implementation. Am J Community Psychol. 2008 Jun;41(3-4):327-50. doi: 10.1007/s10464-008-9165-0. PMID 18322790
- [Background] Weiner BJ. A theory of organizational readiness for change. Implement Sci. 2009 Oct 19;4:67. doi: 10.1186/1748-5908-4-67. PMID 19840381
- [Background] Subedi R, Aitken N, Greenberg L. Canadian Social Environment Typology User Guide. Ottawa, ON: Statistics Canada; 2022.
- [Background] Scaccia JP, Cook BS, Lamont A, Wandersman A, Castellow J, Katz J, Beidas RS. A practical implementation science heuristic for organizational readiness: R = MC2. J Community Psychol. 2015 Apr;43(4):484-501. doi: 10.1002/jcop.21698. Epub 2015 Apr 13. PMID 26668443
- [Background] Miller CJ, Barnett ML, Baumann AA, Gutner CA, Wiltsey-Stirman S. The FRAME-IS: a framework for documenting modifications to implementation strategies in healthcare. Implement Sci. 2021 Apr 7;16(1):36. doi: 10.1186/s13012-021-01105-3. PMID 33827716
- [Background] Wiltsey Stirman S, Baumann AA, Miller CJ. The FRAME: an expanded framework for reporting adaptations and modifications to evidence-based interventions. Implement Sci. 2019 Jun 6;14(1):58. doi: 10.1186/s13012-019-0898-y. PMID 31171014
- [Background] Xie F, Pullenayegum E, Gaebel K, Bansback N, Bryan S, Ohinmaa A, Poissant L, Johnson JA; Canadian EQ-5D-5L Valuation Study Group. A Time Trade-off-derived Value Set of the EQ-5D-5L for Canada. Med Care. 2016 Jan;54(1):98-105. doi: 10.1097/MLR.0000000000000447. PMID 26492214
- [Background] Herdman M, Gudex C, Lloyd A, Janssen M, Kind P, Parkin D, Bonsel G, Badia X. Development and preliminary testing of the new five-level version of EQ-5D (EQ-5D-5L). Qual Life Res. 2011 Dec;20(10):1727-36. doi: 10.1007/s11136-011-9903-x. Epub 2011 Apr 9. PMID 21479777
- See also: Choose to Move website — http://choosetomove.ca
- See also: Active Aging Research Team website — http://activeagingrt.ca